CLINICAL TRIAL: NCT05272956
Title: Impact of Parental Involvement in Enteral Nutrition on Their Presence in Neonatal Units
Brief Title: Parental Involvement in Enteral Nutrition in Neonatal Units
Acronym: PREMALIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 87RI21_0030 (PREMALIM)
Record Dates: First submitted 2022-02-09; First posted 2022-03-10 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Enteral feeding is carried out with a syringe pump
- intervention group (Experimental): the first enteral feeding is pushed with a syringe by the nurse. Following enteral feeding attempts are pushed with a syringe by the parents. Bolus feeding speed is at the discretion of the person pushing the syringe (nurse or parent) and is adjusted to the child's signs of discomfort. When the parents are absent, enteral feeding is carried out with a syringe pump
  Interventions: Procedure: enteral feeding with pushed syringe by the parents

INTERVENTIONS:
Procedure: enteral feeding with pushed syringe by the parents — enteral feeding pushed by parents with a syringe
  Arms: intervention group

SUMMARY:
* Hypothesis : Bolus feeding of the newborn with a syringe under parents' visual control increases parental presence when compared to enteral feeding with a syringe pump.
* Main criteria : Comparison of parental presence (mean time in hours) between the two arms : pushed bolus syringe feeding under parent's visual control and enteral feeding with a syringe pump.

DETAILED DESCRIPTION:
* Nutrition is the cornerstone of neonatology. Adequate nutrition is necessary for a healthy brain growth and a physiological development. When oral feeding skills are not acquired, enteral feeding is used via a nasogastric tube by an electric syringe pump. The birth a premature child jeopardizes parent-infant bonding and hinders parental feeding skills. Family-centered care has shown to be beneficial for the child and his parents by promoting early interactions, which lay the foundations for the child's psychological development. As such, pushed bolus enteral feeding by the parents with a syringe has been a common practice in Sweden since the 1980s to involve the parents in enteral feeding practices. In France, this practice has been used in neonatal intensive care units (NICU). Two French studies on this subject have been published. One focused on using parental pushed bolus enteral feeding in a hospitalization at home setting, whereas the other study investigated the impact of parental observation on pushed bolus enteral feeding. To our knowledge, there is no study proving the superiority of bolus feeding with a syringe under parents' visual control over enteral feeding with a syringe pump.
* This study is an open-label, randomized, comparative interventional study with an intention-to-treat analysis. We compared a control group (enteral nutrition with an electric syringe pump while the neonate is lying in a cocoon or carried by their parent) to an intervention group (pushed bolus enteral nutrition under parents' visual control)
* In the control group, enteral feeding used an electric syringe pump.
* In the intervention group, the first enteral feeding is pushed with a syringe by the nurse. Following enteral feeding attempts are pushed with a syringe by the parents only if they can or will grow. Bolus feeding speed is at the discretion of the person pushing the syringe (nurse or parent) and is adjusted to the child's signs of discomfort. When the parents are absent, enteral feeding is carried out with a syringe pump.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 30 and 34 WA (weeks of amenorrhea)
* Patient affiliated to a social security scheme
* Hospitalized in neonatal intensive care unit (NICU)
* 3 days of life or more

Exclusion Criteria:

Corrected age> 34WA and 4 days

* Mechanical ventilation or non-invasive ventilation with FIO2> 35%
* Serious congenital malformation
* Planned transfer to another hospital
* Enteral nutrition <40ml / kg / day
* Immediate post-operative care
* Multiple pregnancy
* Poor understanding of french

  • Secondary exclusion criteria
* Digestive rest greater than 5 days
* Death
* No enteral nutrition pushed by parents

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
parental presence | from start to the end of enteral feeding, with a maximum of 10 weeks
  Comparison of parental presence (mean time in hours) between the two arms: pushed bolus syringe feeding under parent's visual control and enteral feeding with a syringe pump

SECONDARY OUTCOMES:
Corrected age at which oral feeding skills are acquired | from start to the end of enteral feeding, with a maximum of 10 weeks
  Comparison of corrected age at which oral feeding skill are acquired between the two arms : pushed bolus syringe feeding under parent's visual control and enteral feeding with a syringe pump
Weight gain in g / kg / day during the study time | from start to the end of enteral feeding, with a maximum of 10 weeks
  Comparison of weight gain during the study time between the two arms : pushed bolus syringe feeding under parent's visual control and enteral feeding with a syringe pump
Mean daily skin-to-skin duration | from start to the end of enteral feeding, with a maximum of 10 weeks
  Comparison of mean daily skin-to-skin during the study time between the two arms : pushed bolus syringe feeding under parent's visual control and enteral feeding with a syringe pump
Percentage of breastfeeding at inclusion and at the end of the participation period | from start to the end of enteral feeding, with a maximum of 10 weeks
  Comparison of rate of breastfeeding at inclusion and at the end of the participation period between the two arms : pushed bolus syringe feeding under parent's visual control and enteral feeding with a syringe pump
Anxiety mean score for both parents (PARENTAL STRESSOR SCALE) | from start to the end of enteral feeding, with a maximum of 10 weeks
  Comparison of anxiety level for both parents during the study time between the two arms : pushed bolus syringe feeding under parent's visual control and enteral feeding with a syringe pump. The Parental Stressor Scale (PSS) was published by Margaret S. Miles to evaluate the parental anxiety in neonatal intensive care unit. Higher score is associated with a high level of parental anxiety.
Mother-newborn bond assessment scale (MIBS) score | from start to the end of enteral feeding, with a maximum of 10 weeks
  Comparison of mother-newborn bond assessment between the two arms : pushed bolus syringe feeding under parent's visual control and enteral feeding with a syringe pump.
  The mother-to-infant Bonding Scale (MIBS) published by Taylor in 2005, is a simple 8 item self-rating mother-to-infant bonding questionnaire to assess the feelings of a mother towards her new baby.
Adherence of pushed bolus syringue feeding under parent's visual control | from start to the end of enteral feeding, with a maximum of 10 weeks
  Likert Scale used to evaluate the satisfaction of both parent in pushed bolus syringue feeding under parent's visual control.
  Likert scale provides five possible answers to a statement or question that allows respondents to indicate their positive-to-negative strength of agreement or strength of feeling regarding the question or statement.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Henri Duffaut, Avignon
  - Limoges university hospital, Limoges

IPD SHARING:
Plan to Share IPD: No